CLINICAL TRIAL: NCT02064530
Title: Postoperative Analgesic Effects of Dexmedetomidine Added to Bupivacaine for Transversus Abdominis Plane Block for Lower Abdominal Surgery
Brief Title: Postoperative Analgesic Effects of Dexmedetomidine for Transversus Abdominis Plane Block
Acronym: TAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Recep Aksu, associated prof., TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014/37
Record Dates: First submitted 2014-02-14; First posted 2014-02-17 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-09

CONDITIONS: Pain
Keywords: TAP block; dexmedetomidine; bupivacaine; postoperative analgesia
MeSH Terms: conditions — Pain | interventions — Bupivacaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- bupivacaine (Active Comparator): 0,5% 20 ml bupivacaine added 0.9% 1 ml serum physiologic on TAP block
  Interventions: Drug: Bupivacaine
- dexmedetomidine (Active Comparator): 100 mcg dexmedetomidine added to 0,5% 20 ml bupivacaine on TAP block
  Interventions: Drug: Dexmedetomidine
- serum phsyologic (Sham Comparator): 0,9% 21 ml serum physiologic
  Interventions: Drug: serum physiologic

INTERVENTIONS:
Drug: Bupivacaine — 21 ml 0.5 %bupivacaine is applied interfasially
  Other Names: marcaine
  Arms: bupivacaine
Drug: Dexmedetomidine — 1 ml dexmedetomidin + 20 ml 0.5 % bupivacaine are applied interfasially
  Other Names: precedex
  Arms: dexmedetomidine
Drug: serum physiologic — 21 ml serum physiologic is applied interfasially
  Arms: serum phsyologic

SUMMARY:
the aim of this study is evaluate postoperative analgesic effects of dexmedetomidine added to bupivacaine on TAP block in patients undergoing lower abdominal surgery.

DETAILED DESCRIPTION:
TAP block is being used a method of multimodal balanced analgesia reduces postoperative pain, opioid requirement after surgery and adverse effect of opioid such as sedation, nausea vomiting and ileus. Dexmedetomidine ,an alfa-2 adrenoreceptor agonist, is being used and adjuvant capable of prolonging duration of sensory and motor block on nerve blocks.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2
* 18-65 aged
* patient undergoing lower abdominal surgery

Exclusion Criteria:

* chronic opioid consumption
* bupivacaine and dexmedetomidine allergies
* coagulopathy
* infection at the needle insertion side
* chronic liver and kidney disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
opioid consumption | postoperative 1 day
  patient controlled analgesia

SECONDARY OUTCOMES:
visual analog scale | postoperative 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Recep Aksu, assoc. prof., Study Director — Erciyes universty medicine faculty; Gülçin Patmano, resident, Principal Investigator — Erciyes universty medicine faculty
Locations (1):
- Erciyes universty, Kayseri, Melikgazi, Turkey (Türkiye)